CLINICAL TRIAL: NCT03126500
Title: Post-Hospital Syndrome: Evaluation of Functional Status in Malnourished, Geriatric Patients at Hospital Discharge
Brief Title: Post - Hospital Syndrome: Profile of Functional Status by Malnutrition
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Kristina Norman, PD Dr., Charite University, Berlin, Germany
Other Study IDs: POSTHOSP
Record Dates: First submitted 2017-04-12; First posted 2017-04-24 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Malnutrition; Sarcopenia
Keywords: Malnutrition; Disease-related malnutrition; Frailty; Sarcopenia; Hospital discharge; Geriatrics
MeSH Terms: conditions — Malnutrition; Sarcopenia; Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Malnourished: malnourished, geriatrics patients at hospital discharge

SUMMARY:
Malnutrition is common problem in hospitalized geriatrics at discharge. Malnutrition is a high risk for functional limitations, impaired muscle strength and reduced quality of life.

DETAILED DESCRIPTION:
The majority of geriatric hospitalized patients are at high risk for malnutrition at discharge, which has negative impact on post-hospital outcomes. In a cross-sectional analysis in malnourished, geriatric patients we will evaluate frailty-status and functional status using objective and subjective methods at hospital discharge. Moreover, we will investigate the association between nutritional Status and frailty, sarcopenia, quality of life and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Informed written consent
* Existing or risk of malnutrition
* Normal cognitive status according to Mini-Mental State Examination (MMSE ≥ 24 points)
* Life expectancy of > 3 months according to treating doctor

Exclusion Criteria:

* Age < 60 years
* Lack of informed written consent
* No risk of malnutrition
* Low cognitive status according to Mini-Mental State Examination (MMSE < 24 points)
* Life expectancy of < 3 months according to treating doctor

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants are assessed upon discharge from the hospital. Only malnourished patients were analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-05-31 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Functional Parameter: gait speed | Baseline (hospital discharge)
  gait analysis

SECONDARY OUTCOMES:
Functional Parameter: timed up & go (TUG) time | Baseline (hospital discharge)
  timed up & go (TUG) test
Functional Parameter: stair climbing time | Baseline (hospital discharge)
  stair climbing test
Functional Parameter: Peak expiratory flow rate | Baseline (hospital discharge)
  peak flow meters scale
Strength Parameter: Hand grip strength | Baseline (hospital discharge)
  Hand grip strength measurement
Strength Parameter: Knee extension strength | Baseline (hospital discharge)
  Knee extension strength measurement
Index of quality of life | Baseline (hospital discharge)
  validated questionnaire
Body composition | Baseline (hospital discharge)
  bioelectric impedance Analysis
Frailty-Status | Baseline (hospital discharge)
  Fried criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University, Berlin, Germany, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No